CLINICAL TRIAL: NCT06447701
Title: Effect of Interleukin-6 Receptor Inhibition for Avoiding Recurrence of Ischemic Stroke in Patients With Symptomatic Intracranial Atherosclerosis: a Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Interleukin-6 Receptor Inhibition for Symptomatic Intracranial Atherosclerosis
Acronym: IRIS-sICAS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Collaborators: Shenzhen Second People's Hospital (Other); Central People's Hospital of Zhanjiang (Other); Shantou Central Hospital (Other); Eighth Affiliated Hospital, Sun Yat-sen University (Other); Guangzhou First People's Hospital (Other); Peking University Shenzhen Hospital (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LC2024ZD025
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Brain Diseases; Ischemic Stroke; Ischemia; Stroke; Cerebral Infarction; Atherosclerosis of Artery; Atheroscleroses, Intracranial
Keywords: Tocilizumab; Symptomatic intracranial atherosclerotic stenosis; Recurrence; Ischemic stroke
MeSH Terms: conditions — Brain Diseases; Ischemic Stroke; Ischemia; Stroke; Cerebral Infarction; Intracranial Arteriosclerosis; Recurrence | interventions — tocilizumab

STUDY DESIGN:
Intervention Model Description: The subject numbers and corresponding medication numbers are permanently identified and unique for each successfully randomized patient. If any patients who have been successfully randomized do not receive the trial medication or cannot be reassigned to others, their medication and medication numbers will be invalidated by the medication administrator. To ensure blinding during the trial execution, unblinded personnel responsible for administering and configuring the trial drug must sign a confidentiality agreement. Investigators, other blinded investigators, subjects, and sponsors will not have access to any information regarding group assignment or related documents pertaining to the trial drug.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The subject numbers and corresponding medication numbers are permanently identified and unique for each successfully randomized patient. If any patients who have been successfully randomized do not receive the trial medication or cannot be reassigned to others, their medication and medication numbers will be invalidated by the medication administrator. To ensure blinding during the trial execution, unblinded personnel responsible for administering and configuring the trial drug must sign a confidentiality agreement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tocilizumab group (Experimental): Intravenously for more than 1 hour.
  Interventions: Drug: Tocilizumab
- Control group (Placebo Comparator): Intravenously for more than 1 hour.
  Interventions: Drug: NaCl 0.9% 100ml

INTERVENTIONS:
Drug: Tocilizumab — Single dose intravenous application
  Arms: Tocilizumab group
Drug: NaCl 0.9% 100ml — Single dose intravenous application
  Arms: Control group

SUMMARY:
IRIS-sICAS is a multicenter, randomized, double-blind, placebo-controlled clinical trialis a multicenter, randomized, double-blind, placebo-controlled clinical trial, to assess the safety and efficacy of tocilizumab injection in lowering the incidence of newly diagnosis ischemic stroke and improving prognosis in symptomatic intracranial atherosclerosis patients.

DETAILED DESCRIPTION:
Intracranial atherosclerosis (ICAS) is one of the most common causes of stroke worldwide, and the currently recommended intensive pharmacologic and surgical treatments show only modest efficacy, with approximately 20% of strokes still recurring, for which there is no targeted treatment. Tocilizumab is a recombinant humanized anti-human interleukin-6 receptor monoclonal antibody that exerts anti-inflammatory effects by specifically binding to the IL-6 receptor and blocking IL-6 signal transduction. Previous studies have shown that tocilizumab can effectively attenuate acute ischemic injury in the early stage of myocardial infarction and has potentially anti-atherosclerotic effects. However, application in ICAS not yet reported. This study is a multicenter, randomized, double-blind, placebo-controlled clinical trial, which enrolled patients with symptomatic ICAS occurring within 72 hours of ischemic stroke or high-risk transient ischemic attack. Patients who consented to participate in the study were randomly assigned in a 1:1 ratio to receive a single infusion of 320mg tocilizumab or placebo (saline injection), and patients were followed up to assess the safety and efficacy of tocilizumab injection in lowering the incidence of newly diagnosis ischemic stroke and improving prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant women with acute stroke symptoms aged over 18 years.
* Patients having an ischemic stroke or a TIA prior to randomization (Patients having an acute ischemic stroke within 72 hours with NIHSS score≤5 at baseline, or patients having a TIA within 72 hours with Oxfordshire Community Stroke Project on the basis of age, blood pressure, clinical features, and duration of TIA symptoms (ABCD2) score≥4 at baseline).
* The entry event is attributed to symptomatic atherosclerosis (50-99%) in an intracranial qualifying artery (intracranial carotid artery (C4-7), middle cerebral artery (M1), intracranial vertebral artery or basilar artery) confirmed by CT, MR angiography, or digital subtraction angiography.
* Informed consent obtained from patients or their legal representatives.
* Willing to be followed up as required by the clinical study protocol.

Exclusion Criteria:

* Thrombolytic therapy or thrombectomy within 24 hours prior to enrollment.
* Pre-stroke mRS score ≥ 2.
* Combined or previous intracranial hemorrhage: hemorrhagic stroke, epidural hematoma, subdural hematoma, intraventricular hemorrhage, subarachnoid hemorrhage, etc.
* Any of the following unequivocal cardiac source of embolism: chronic or paroxysmal atrial fibrillation, sinus node dysfunction, mitral stenosis, prosthetic heart valves, endocarditis, left ventricular mural thrombus or valvular vegetation, myocardial infarction within three months, dilated cardiomyopathy, spontaneous echogenic defects in the left atrium or an ejection fraction of less than 30%.
* Intracranial arterial stenosis due to arterial dissection, Moya Moya disease; herpes zoster, varicella zoster or other viral vasculopathy; neurosyphilis; radiation induced vasculopathy; fibromuscular dysplasia; sickle cell disease; neurofibromatosis; post-partum angiopathy; suspected vasospastic process, suspected recanalized embolus; any known vasculitic disease.
* Extracranial stenosis ≥50%, subclavian arterial stenosis≥50% or subclavian steal syndrome.
* Previous interventions for intracranial arterial stenosis.
* Concurrent intracranial tumors, intracranial aneurysms or arteriovenous malformations
* Neutrophil < 2×10 9/L.
* Platelet < 100×10 9/L.
* Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) levels greater than 1.5 times the upper limit of normal.
* Active infections including localized.
* Evidence of HIV or hepatitis B positivity.
* Positive tuberculosis-related tests.
* Concurrent peptic ulcer, diverticulitis or inflammatory bowel disease.
* Concurrent malignant tumors, recent bone marrow transplant or recent organ transplant.
* Systolic blood pressure ≥ 180 mmHg or diastolic blood pressure ≥ 110 mmHg despite blood pressure control.
* Known allergy to tocilizumab or excipients.
* Use of immunosuppressive drugs or systemic use of antibiotics.
* Received any live or live attenuated vaccine within 4 weeks prior to enrollment or plan to receive a live or live attenuated vaccine during the study.
* History of demyelination or presence of neurological symptoms suggestive of demyelination.
* Previously existing neurological or psychiatric disorders that could potentially confuse neurological function assessment.
* An expected survival less than 90 days.
* Participation in another interventional clinical study.
* Patients unsuitable for enrollment in the clinical trial according to investigators decision making.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 486 (Estimated)
Dates: Start 2025-10-30 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with newly diagnosed ischemic stroke within 90(±7) days | 90(±7) days
  Stroke is defined as an acute episode of focal neurological dysfunction associated with cerebral vascular injury, with no apparent non-vascular cause such as brain infection, trauma, tumor, seizure, severe metabolic disease, or degenerative neurological disease.
  Ischemic stroke is defined as an acute episode of a new focal neurological deficit lasting >24 hours, an increase in existing focal neurological deficit lasting >24 hours, or a focal neurological deficit lasting <24 hours that is associated with evidence of new ischemic changes based on neuroimaging. The focal neurological deficit is not attributable to a non-ischemic etiology. Hemorrhage may be a consequence of ischemic stroke, and in this situation, the stroke is an ischemic stroke with hemorrhagic transformation but not a hemorrhagic stroke.

SECONDARY OUTCOMES:
The functional neurological status at 6(±1) days or discharge if earlier from baseline | 6(±1) days
  The functional neurological status is evaluated through National Institute of Health Stroke Scale(NIHSS). The NIHSS is a standardized neurological examination score that is a valid and reliable measure of disability and recovery after acute stroke. Scores range from 0 to 42, with higher scores indicating more severe disability. The scale includes measures of level of consciousness, extra ocular movements, motor and sensory tests, coordination, language and speech evaluations.
The incidence of composite events including any type of stroke (ischemic stroke(IS), subarachnoid hemorrhage(SAH), or intracerebral hemorrhage(ICH)), myocardial infarction(MI), and transient ischemic attack(TIA) and each of foresaid events at 30(±3) days | 30(±3) days
  IS is defined as an acute episode of a new focal neurological deficit lasting >24 hrs, an increase in existing focal neurological deficit lasting >24 hrs, or a focal neurological deficit lasting <24 hrs that is associated with evidence of new ischemic changes based on neuroimaging. The focal neurological deficit is unrelated to a non-ischemic etiology. Hemorrhage may be a result of IS.
  Hemorrhagic stroke including SAH and ICH is defined as a new focal neurological deficit caused by a nontraumatic intraparenchymal hemorrhage, with neuroimaging evidence of corresponding intraparenchymal hemorrhage, except hemorrhagic transformation of an IS.
  MI is defined as an episode of myocardial necrosis in a clinical setting consistent with myocardial ischemia.
  TIA is defined as a transient episode of a focal ischemic neurological deficit resolving completely within 24 hrs, caused by focal cerebral or retinal ischemia, without evidence of corresponding cerebral infarction based on neuroimaging.
The incidence of composite events including any type of stroke (ischemic stroke(IS), subarachnoid hemorrhage(SAH), or intracerebral hemorrhage(ICH)), myocardial infarction(MI), and transient ischemic attack(TIA) and each of foresaid events at 90(±7) days | 90(±7) days
  IS is defined as an acute episode of a new focal neurological deficit lasting >24 hrs, an increase in existing focal neurological deficit lasting >24 hrs, or a focal neurological deficit lasting <24 hrs that is associated with evidence of new ischemic changes based on neuroimaging. The focal neurological deficit is unrelated to a non-ischemic etiology. Hemorrhage may be a result of IS.
  Hemorrhagic stroke including SAH and ICH is defined as a new focal neurological deficit caused by a nontraumatic intraparenchymal hemorrhage, with neuroimaging evidence of corresponding intraparenchymal hemorrhage, except hemorrhagic transformation of an IS.
  MI is defined as an episode of myocardial necrosis in a clinical setting consistent with myocardial ischemia.
  TIA is defined as a transient episode of a focal ischemic neurological deficit resolving completely within 24 hrs, caused by focal cerebral or retinal ischemia, without evidence of corresponding cerebral infarction based on neuroimaging.
Proportion of patients with functional independence at 90(±7) days | 90(±7) days
  Functional independence is defined as the modified Rankin Scale(mRS) score ranging from 0-2.
  The mRS is a valid and reliable clinician-reported measure of global disability that has been widely applied for evaluating recovery from stroke. It is a scale used to measure functional recovery (the degree of disability or dependence in daily activities) of people who have suffered a stroke. mRS scores range from 0 to 6, with 0 indicating no residual symptoms; 5 indicating bedbound, requiring constant care; and 6 indicating death.
Health-related quality of life at 90(±7) days | 90(±7) days
  Health-related quality of life is assessed with the European Quality Five Dimensions Five Level scale (EQ-5D-5L).
  The EQ-5D-5L is a generic instrument for describing and valuing health. It is based on a descriptive system that defines health in terms of five dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. Each dimension has five response categories corresponding to: no problems, slight, moderate, severe and extreme problems. The instrument is designed for self-completion, and respondents also rate their overall health on the day of the interview on a 0-100 hash-marked, vertical visual analogue scale.
Mortality at 90(±7) days | 90(±7) days
  Mortality rates are defined as the number of deaths observed divided by the number of subjects observed over the 90-day study period.
Incidence of serious adverse events | 90(±7) days
  Including but not limited to acute respiratory failure, severe or malignant cerebral artery infarction, acute heart failure, debridement decompression, and other major medical events that can result in death, immediately life-threatening, hospitalization or prolongation of this hospitalization, terminally or severely disabling/incapacitating, the loss of a significant ability to maintain normal life functioning, or medical intervention to avoid the above outcomes.
Change of inflammatory blood biomarkers from admission to 72 hours | 72 hours
  Interleukin-6 (IL-6)
Change of inflammatory blood biomarkers from admission to 72 hours | 72 hours
  hypersensitive C-reactive protein (hsCRP)

IPD SHARING:
Plan to Share IPD: No